CLINICAL TRIAL: NCT04198246
Title: The Chinese Essential Tremor Registry
Brief Title: Chinese ET Registry (CETR)
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CETR
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Essential Tremor
Keywords: Motor symptoms; Nonmotor symptoms; Natural history; The Essential Tremor Rating Assessment Scale (TETRAS)
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extraction of DNA from peripheral blood of patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese Essential Tremor Registry (CETR) is to develop a database of patients with Essential tremor in China.

DETAILED DESCRIPTION:
Essential tremor (ET) is one of the most common movement disorders and affects approximately 1% of the population worldwide. Twin and family history studies show a high heritability for essential tremor. The molecular genetic determinants of essential tremor are unknown. Some mutations have been found in ET families but have not been validated in others. The pathophysiological basis of ET remains unknown. In 2017, a task force of the International Parkinson and Movement Disorder Society proposed a new formal definition of essential tremor as a syndrome of isolated tremor of both upper limbs with a duration of at least 3 years, with or without tremor in other locations, such as head, larynx (voice tremor), or lower limbs. Defining essential tremor as a syndrome and not as a single disease, while concomitantly narrowing its phenotypic scope to increase its homogeneity, recognizes that there are multiple possible causes, which may facilitate progress in understanding the pathogenesis. Investigators aim to establish a database of longitudinal recruited ET cohort, and characterize the clinical feature, genetic basis, environmental factors and their interactions among different ET subtypes in China, identify natural history of a highly-presentative Chinese ET cohort and to discern major milestones in the disease process which indicates disease progression.

Data were collected at baseline. Information about detailed disease history, level of education, significant chronic comorbidities, physical examination, medication history, family history, living habits and toxic exposure history, which include smoking, drinking tea, alcoholic consumption, drinking coffee, exposure to pesticide or occupational solvent, history of carbon monoxide poisoning and recurrent head trauma will be recorded at baseline. For each evaluation, the same questionnaires will be conducted. A standardized neurological assessment according to the recommendation of Consensus on the construction of clinical database of Parkinson's disease and movement disorders in China.

The Essential Tremor Rating Assessment Scale (TETRAS) includes both performance and Activities of Daily Living (ADL) subscales. It is conducted for the clinical measurement of ET severity and tremor's impact on ADL. The non-motor symptoms are evaluated by Non-motor Symptom Scale (NMSS).Functional constipation was diagnosed by the Rome III diagnostic criteria. Excessive daytime sleepiness was evaluated by Epworth Sleepiness Scale (ESS). Probable rapid eye movement sleep behavior disorder (p-RBD) was diagnosed by rapid eye movement sleep behavior questionnaire-Hongkong (RBDQ-HK). Restless leg syndrome (RLS) was diagnosed with the Cambridge Hopkins Restless Leg syndrome questionnaire (CH-RLSq). Cognitive assessment was used the previously validated scale, Mini Mental State Examination (MMSE). Olfaction test was carried out by Hyposmia Rating Scale (HRS), a proportion of patients was also ascertained by Sniffin's Sticks. Depression was diagnosed by Hamilton Depression Scale (HAMD).DNA samples extracted from peripheral blood and all the ET patients will be examed by Whole Exome Sequencing or Whole-genome sequencing. All the participants are scanned by structural MRI to exclude obvious intracranial lesions and other metabolic disorders, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ET by the Consensus Statement on the Classification of Tremors,From the Task Force on Tremor of the International Parkinson and Movement Disorder Society.

Exclusion Criteria:

* Lack of capacity to consent to participate in the project.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Most of the ET patients comes from mainland China, especially from Hunan Province, Hubei Province, Jiangxi Province and Guizhou Province. The proportion of male patients is slightly dominant than that of female patients. The age of ET patients ranges from 13 to more than 90 years old.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The tremor's impact on activities of daily living and clinical measurement of ET severity are evaluated by The Essential Tremor Rating Assessment Scale (TETRAS). | baseline
  TETRAS consists of two subscales. The first one, Activities of Daily Living (ADL) Subscale contains 12 self-scored items, rating tremor's impact on ADL in a 0-4 Likert-type scale. Total score varies from 0-48. Higher score indicates a bigger impact on activities of daily living. The second part is the Performance Subscale, and is rated by clinicians'examination. The subscale is formed by 9 items that rate action tremor in the head, face, voice, limbs, and trunk from 0 to 4. Total score varies from 0-64. Higher score indicates severer tremor. For most items, the scores are defined only by whole numbers, but 0.5 increments may be used if you believe the rating is between two whole number ratings and cannot be reconciled to a whole number. Each 0.5 increment in rating is specifically defined for the assessment of upper limb postural and kinetic tremor and the dot approximation task (items 4 and 8).
The non-motor symptoms are evaluated by Non-motor Symptom Scale. | baseline
  This scale includes 30 items which is divided into 9 domains. Total score varies from 0-360. Higher score indicates severer symptoms. Domain 1 evaluates cardiovascular system symptoms. Score of domain 1 varies from 0-24. Domain 2 evaluates sleep condition. Score of domain 2 varies from 0-48. Domain 3 evaluates cognitive function. Score of domain 3 varies from 0-72. Domain 4 evaluates illusion. Score of domain 4 varies from 0-36. Domain 5 evaluates attention and memory. Score of domain 5 varies from 0-36. Domain 6 evaluates gastrointestinal symptoms. Score of domain 6 varies from 0-36. Domain 7 evaluates urinary symptoms. Score of domain 7 varies from 0-36. Domain 8 evaluate sensory symptoms. Score of domain 8 varies from 0-24. Domain 9 evaluates other non-motor symptoms. Score of domain 9 varies from 0-48.
Cognitive condition is assessed by Mini Mental State Examination. | baseline
  This scale includes 30 items. Score of all the questions will be summed. All items were rated on a 2-point scale (0-1), with a minimal score of 0, and maximum total score of 30. A higher score demonstrates more better cognitive condition. The definition of cognitive disorder differs in education level. For illiteracy, presence of cognitive impairment is defined as MMSE score. For those only receive elementary education, the cut-off value is 20. For other patients, presence of cognitive impairment was defined as MMSE scores less than 25.
Olfaction test was measured by Hyposmia Rating Scale. | baseline
  This scale includes 6 items. Score of all the questions will be summed. All items were rated on a 4-point scale (1-4), with a minimal score of 6, and maximum total score of 24. A higher score demonstrates more worse sense of olfaction. The cutoff value HRS is 22.5.
Depression was diagnosed by Hamilton and Montgomery-Asberg Depression Scale. | baseline
  This scale includes 17 items. Score of all the questions will be summed. Total score ranges from0-53. A higher score demonstrates more severer depression. The study participants were defined to be not depressed (scores 0-6), to have minor depression (scores 7-14), or to have major depression (scores above 14) at the different visits during follow-up.

SECONDARY OUTCOMES:
Constipation was diagnosed by Functional Constipation Diagnostic Criteria Rome III. | baseline
  The diagnostic criteria must include two or more of the following:
  1. Straining during at least 25% of defecations
  2. Lumpy or hard stools in at least 25% of defecations
  3. Sensation of incomplete evacuation for at least 25% of defecations
  4. Sensation of anorectal obstruction/blockage for at least 25% of defecations
  5. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
  6. Fewer than three defecations per week 2. Loose stools are rarely present without the use of laxatives 3.
  Insufficient criteria for irritable bowel syndrome * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
Excessive sleepiness is evaluated by Epworth Sleepiness Scale. | baseline
  This scale includes 8 items. Score of all the questions will be summed. All items were rated on a 4-point scale (0-3), with a minimal score of 0, and maximum total score of 24. A higher score demonstrates more severe excessive daytime sleepiness. Participants were classified as showing excessive daytime sleepiness if their total score ≥10.
Probable rapid eye movement sleep behavior disorder was diagnosed by Probable rapid eye movement sleep behavior disorder Questionnaire-Hongkong. | baseline
  This scale includes 13 items. Score of all the questions will be summed. Total score of the answers ranges from 0 to 100, where higher scores reflect severer rapid eye movement sleep behavior disorder. The optimal cutoff value for the overall scale is 17; subjects were classified as showing RBD when they reached the above score.
Restless leg syndrome (RLS) was diagnosed with the Cambridge Hopkins Restless Leg syndrome questionnaire. | baseline
  1. have, or have you had, recurrent uncomfortable feelings or sensations in your legs while you are sitting or lying down
  2. have, or have you had, a recurrent need or urge to move your legs while you were sitting or lying down
  3. more likely to have these feelings when you are resting
  4. If you get up or move around when you have these feelings, these feelings get better
  5. these feelings in your legs most likely to occur at mid-day or afternoon or evening or night
  6. Simply changing leg position by itself once without continuing to move usually relieve these feelings usually don't relieves
  7. These feelings are not or not always due to muscle cramps

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China